CLINICAL TRIAL: NCT02360631
Title: Advancing Tobacco Use Treatment for African American Smokers
Acronym: KIS-IV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lisa Sanderson Cox, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Lisa Sanderson Cox, PhD, Research Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000721; R01DA035796 (NIH)
Record Dates: First submitted 2015-02-04; First posted 2015-02-10 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Smoking Cessation
Keywords: smoking; quit smoking; smoking treatment
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chantix (varenicline) (Experimental): Participants will receive 1mg pills to take twice a day for 12 weeks.
  Interventions: Drug: Chantix
- Placebo (Placebo Comparator): Participants will receive a placebo pill to take twice a day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chantix — A drug used to treat nicotine addiction.Chantix is approved by the FDA to be given to help people quit smoking.
  Other Names: Varenicline
  Arms: Chantix (varenicline)
Drug: Placebo — Health education counseling will be provided to all participants.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether or not providing Chantix (varenicline) will help African American smokers quit smoking.

DETAILED DESCRIPTION:
To have an impact on the premature mortality of African American smokers, effective treatment for smokers across the smoking continuum must be identified. Varenicline, the leading first-line medication for tobacco use treatment, triples the likelihood of long-term abstinence relative to placebo in those smoking >10 cpd. To date, efficacy of varenicline has not been established in African American smokers or light smokers. The long-term goal of this research is to advance treatment for all African American smokers in order to reduce tobacco-related disease and death. Our primary objective is to evaluate the efficacy of varenicline for tobacco use treatment among 500 African American smokers, including a full range of cpd, within a double-blind, placebo-controlled, randomized clinical trial. We will randomize participants in a 3:2 ratio to receive varenicline (1 mg bid; n=300) or placebo (n=200) for 12 weeks, along with individualized health education counseling for all participants. Our specific aims are to evaluate the efficacy of varenicline to promote abstinence in African American smokers across the continuum of smoking level, to examine efficacy in light smokers and also in moderate to heavy smokers, and to describe biopsychosocial characteristics of this group and evaluate in relation to abstinence. This innovative study will provide the first placebo-controlled evaluation of varenicline in the full spectrum of African American smokers, and the first to examine varenicline in light smokers. Findings will contribute to advancing effective treatment for African American smokers and for light smokers, and enhancing individualized treatment. Increased treatment efficacy will have major impact on reducing tobacco-related morbidity and mortality in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African American
* Smokes ≥ 1 cigarette per day (cpd)
* Smoke on ≥ 25 days of the past 30 days
* Functioning telephone
* Interested in quitting smoking
* Interested in taking 3 months of varenicline
* Willing to complete all study visits

Exclusion Criteria:

* Renal impairment
* Evidence or history of clinically significant allergic reactions to varenicline
* A cardiovascular event in the past month
* History of alcohol or drug dependence in the past year
* Major depressive disorder in the last year requiring treatment
* History of panic disorder, psychosis, bipolar disorder, or eating disorders
* Use of tobacco products other than cigarettes in past 30 days
* Use of pharmacotherapy in the month prior to enrollment, including prior use of varenicline
* Pregnant, contemplating getting pregnant, or breastfeeding
* Plans to move from Kansas City during the treatment and follow-up phase
* Another household member enrolled in the study
* Evidence of current severe major depressive disorder or suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Sanderson Cox, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Swope Health Central, Kansas City, Missouri

REFERENCES:
- [Derived] Lambart L, Nollen NL, Mayo MS, Funk O, Leavens E, Cruvinel E, Brown A, Ahluwalia JS, Sanderson Cox L. The impact of blunt use on smoking abstinence among Black adults: Secondary analysis from randomized controlled smoking cessation clinical trial. Addict Behav. 2024 Jan;148:107877. doi: 10.1016/j.addbeh.2023.107877. Epub 2023 Oct 4. PMID 37804748
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Cox LS, Nollen NL, Mayo MS, Faseru B, Greiner A, Ellerbeck EF, Krebill R, Tyndale RF, Benowitz NL, Ahluwalia JS. Effect of Varenicline Added to Counseling on Smoking Cessation Among African American Daily Smokers: The Kick It at Swope IV Randomized Clinical Trial. JAMA. 2022 Jun 14;327(22):2201-2209. doi: 10.1001/jama.2022.8274. PMID 35699705

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chantix (Varenicline) | Placebo
Started | 300 | 200
Week 12 | 249 | 165
Completed | 267 | 174
Not Completed | 33 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chantix (Varenicline) | Placebo | Total
Number analyzed (Participants) | 300 | 200 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.9) | 52.4 (11.0) | 51.9 (11.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 156 | 106 | 262
  Male | 144 | 94 | 238
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 300 | 200 | 500
Employed [Count of Participants; unit: Participants] | 143 | 113 | 256
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.6 (7.1) | 30.1 (7.6) | 30.4 (7.3)
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 12.9 (6.9) | 12.2 (6.2) | 12.6 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Smoking Abstinence at Month 6
Description: Biochemically verified 7-day point prevalence abstinence defined as smoking zero cigarettes at Month 6 visit
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Chantix (Varenicline) | Placebo
Number analyzed (Participants) | 300 | 200
Participants | 47 | 13

2. Secondary Outcome: Number of Participants With Smoking Abstinence at Week 12
Description: Biochemically verified 7-day point prevalence abstinence defined as smoking zero cigarettes at Week 12 visit
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Chantix (Varenicline) | Placebo
Number analyzed (Participants) | 300 | 200
Participants | 56 | 14

3. Secondary Outcome: Number of Participants With Smoking Abstinence at Week 26
Description: Intent to treat Cotinine verified cessation for light and moderate to heavy smokers by treatment
Time Frame: Week 26
Population: 300 participants received varenicline and of those 154 were Light smokers (10 or less cigarettes per day (CPD) and 146 were moderate to heavy smokers (greater than 10 )CPD. 200 participants received placebo medication and of those 106 were light smokers and 94 were moderate to heavy smokers.
Measure: Count of Participants; unit: Participants
Arm/Group | Chantix (Varenicline) | Placebo
Number analyzed (Participants) | 300 | 200
Participants
  Light: number analyzed (Participants) | 154 | 106
  Light | 33 | 9
  Heavy: number analyzed (Participants) | 146 | 94
  Heavy | 14 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was systematically collected between weeks 0-16.
Arm/Group | Chantix (Varenicline) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/300 | 2/200
Other Adverse Events (participants affected / at risk) | 276/300 | 178/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chantix (Varenicline) (N=300) | Placebo (N=200)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchial inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chantix (Varenicline) (N=300) | Placebo (N=200)
Change in hostility or aggression (Psychiatric disorders) | 99 (99) | 79 (79)
Fatigue or Loss of Energy (General disorders) | 163 (163) | 112 (112)
Nausea (Gastrointestinal disorders) | 163 (163) | 90 (90)
Trouble sleeping (General disorders) | 190 (190) | 117 (117)
Headaches (General disorders) | 157 (157) | 95 (95)
Abnormal dreams (General disorders) | 146 (146) | 93 (93)
Gas or flatulence (Gastrointestinal disorders) | 191 (191) | 130 (130)
Constipation (Gastrointestinal disorders) | 120 (120) | 78 (78)
Dizziness (General disorders) | 95 (95) | 62 (62)
Dry mouth (General disorders) | 183 (183) | 129 (129)
Irritability (Psychiatric disorders) | 167 (167) | 111 (111)

LIMITATIONS AND CAVEATS:
Findings cannot be generalized to non-US Blacks and require replication with smokers outside the Midwestern US.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT02360631/Prot_SAP_000.pdf